CLINICAL TRIAL: NCT00954174
Title: A Randomized Phase III Trial of Paclitaxel Plus Carboplatin Versus Ifosfamide Plus Paclitaxel in Chemotherapy-Naive Patients With Newly Diagnosed Stage I-IV, Persistent or Recurrent Carcinosarcoma (Mixed Mesodermal Tumors) of the Uterus, Fallopian Tube, Peritoneum or Ovary
Brief Title: Paclitaxel and Carboplatin or Ifosfamide in Treating Patients With Newly Diagnosed, Persistent or Recurrent Uterine, Ovarian, Fallopian Tube, or Peritoneal Cavity Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0261; NCI-2011-01959 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000651458; GOG-0261 (Other: NRG Oncology); GOG-0261 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Mixed Mesodermal (Mullerian) Tumor; Ovarian Carcinosarcoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage I Ovarian Cancer AJCC v6 and v7; Stage IA Fallopian Tube Cancer AJCC v6 and v7; Stage IA Ovarian Cancer AJCC v6 and v7; Stage IA Uterine Sarcoma AJCC v7; Stage IB Fallopian Tube Cancer AJCC v6 and v7; Stage IB Ovarian Cancer AJCC v6 and v7; Stage IB Uterine Sarcoma AJCC v7; Stage IC Fallopian Tube Cancer AJCC v6 and v7; Stage IC Ovarian Cancer AJCC v6 and v7; Stage IC Uterine Sarcoma AJCC v7; Stage II Ovarian Cancer AJCC v6 and v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIA Uterine Sarcoma AJCC v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIB Uterine Sarcoma AJCC v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIA Uterine Sarcoma AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIB Uterine Sarcoma AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IIIC Uterine Sarcoma AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7; Stage IVA Uterine Sarcoma AJCC v7; Stage IVB Uterine Sarcoma AJCC v7; Uterine Carcinosarcoma
MeSH Terms: conditions — Carcinosarcoma; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Ifosfamide; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on day 1.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm II (paclitaxel, ifosfamide) (Experimental): Patients receive ifosfamide IV over 1 hour on days 1-3 followed by paclitaxel as in Arm I.
  Interventions: Drug: Ifosfamide; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (paclitaxel, carboplatin)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Arm II (paclitaxel, ifosfamide)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies paclitaxel and carboplatin see how well they work compared with paclitaxel and ifosfamide in treating patients with fallopian tube, or peritoneal cavity cancer that is newly diagnosed, persistent, or has come back (recurrent). Drugs used in chemotherapy, such as paclitaxel, carboplatin, and ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether paclitaxel is more effective when given with carboplatin or ifosfamide in treating patients with uterine, ovarian, fallopian tube, or peritoneal cavity cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if treatment with combination paclitaxel and carboplatin (TC) chemotherapy does not result in an inferior death rate when compared to ifosfamide, mesna, and paclitaxel chemotherapy.

SECONDARY OBJECTIVES:

I. To determine if treatment with combination paclitaxel and carboplatin (TC) chemotherapy does not result in an inferior progression-free survival when compared to ifosfamide, mesna, and paclitaxel chemotherapy.

II. To determine if acute toxicity, specifically physician-assessed neurotoxicity and infection, associated with combination paclitaxel and carboplatin chemotherapy is reduced compared to that of ifosfamide, mesna, and paclitaxel chemotherapy.

III. To determine if treatment with combination paclitaxel and carboplatin chemotherapy is associated with superior patient-reported quality of life and neurotoxicity scores compared to that of ifosfamide, mesna, and paclitaxel chemotherapy.

TERTIARY OBJECTIVES:

I. To bank formalin-fixed, paraffin-embedded (FFPE) tumor tissue and deoxyribonucleic acid (DNA) extracted from whole blood for future research.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours followed by carboplatin IV over 30-60 minutes on day 1.

ARM II: Patients receive ifosfamide IV over 1 hour on days 1-3 followed by paclitaxel as in Arm I.

In both arms, treatment repeats every 21 days for 6-10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed stage I-IV, persistent or recurrent (including unstaged) uterine carcinosarcoma (malignant mixed mullerian tumor-MMMT or with ovarian, fallopian tube or peritoneal carcinosarcoma and an enrollment date prior to 10/21/2013; pathology confirmed by site/institutional pathologist prior to enrollment) and be chemotherapy naïve as directed against their carcinosarcoma; unstaged patients (patients who have not had hysterectomy or ovarian surgery) are eligible and should be included as "unstaged" if the only histologic (pathology) documentation of the disease is a biopsy or curettage of the uterus; if these patients have documented metastatic disease, it should be assigned the appropriate stage (III/IV)
* Patients may have received prior adjuvant external beam radiation therapy and/or vaginal brachytherapy; patients should be at least 4 weeks from the completion of external beam radiotherapy prior to beginning protocol chemotherapy; patients do not need to be delayed if receiving vaginal brachytherapy only
* Gynecologic Oncology Group (GOG) performance status 0, 1, or 2
* Patients must have recovered from the effects of recent surgery, radiotherapy, or other therapy
* Patients must be free of active infection requiring antibiotics
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to beginning protocol chemotherapy; continuation of hormone replacement therapy is permitted
* Platelet count greater than or equal to 100,000/mcL
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL equivalent to Common Terminology Criteria for Adverse Events (CTCAE) version (v)3.0 grade 1
* Creatinine less than or equal to 1.5 times upper limit of normal (ULN), CTCAE v3.0 grade 1
* Bilirubin less than or equal to 1.5 times ULN (CTCAE v3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 times ULN (CTCAE v3.0 grade 1)
* Alkaline phosphatase less than or equal to 2.5 times ULN (CTCAE v3.0 grade 1)
* Serum albumin should be equal to or greater than 3 g/dL
* Neuropathy (sensory and motor) less than or equal to CTCAE v3.0 grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients of childbearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception
* Patients may have measurable disease or non-measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT; measurable disease patients must have at least one "target lesion" to be used to assess progression on this protocol as defined by Response Evaluation Criteria In Solid Tumors (RECIST); tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy

Exclusion Criteria:

* Patients who have received prior cytotoxic chemotherapy for management of uterine or ovarian carcinosarcoma
* Patients with a history of other invasive malignancies or with a concomitant invasive malignancy, with the exception of non-melanoma skin cancer, if there is any evidence of other malignancy being present within the last five years; patients are also ineligible if their previous cancer treatment contraindicates this protocol therapy
* Patients for whom radiotherapy is planned after or during chemotherapy prior to progression of cancer
* Patients with known hypersensitivity to Escherichia (E.) coli-derived drug preparations (pegfilgrastim and filgrastim [G-CSF])
* Patients with a known hypersensitivity to mesna or other thiol compounds
* For enrollment prior to 10/21/2013, patients who are not biopsy proven to have carcinosarcoma of the uterus, fallopian tube, peritoneum or ovary; for enrollment after 10/21/2013, patients who are not biopsy proven to have carcinosarcoma of the uterus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2009-08-17 (Actual); Primary Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Powell, Principal Investigator — NRG Oncology
Locations (538):
- United States (532):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Gynecologic Oncology Associates-Newport Beach, Newport Beach, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Mercy Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- South Korea (6):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul

REFERENCES:
- [Derived] Powell MA, Filiaci VL, Hensley ML, Huang HQ, Moore KN, Tewari KS, Copeland LJ, Secord AA, Mutch DG, Santin A, Warshal DP, Spirtos NM, DiSilvestro PA, Ioffe OB, Miller DS. Randomized Phase III Trial of Paclitaxel and Carboplatin Versus Paclitaxel and Ifosfamide in Patients With Carcinosarcoma of the Uterus or Ovary: An NRG Oncology Trial. J Clin Oncol. 2022 Mar 20;40(9):968-977. doi: 10.1200/JCO.21.02050. Epub 2022 Jan 10. PMID 35007153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 637 subjects were enrolled between 08/17/2009 and 3/24/14. Enrollment initially included uterine carcinosarcoma and was expanded to ovarian carcinosarcoma in June 2010 and then to include fallopian tube and peritoneal carcinosarcoma in October 2013. The primary analysis was restricted to patients with uterine carcinosarcoma.
Groups:
- Regimen I - Uterine Carcinsarcoma Subjects: Paclitaxel 175 mg/m2 IV over 3 hours Day 1. Carboplatin (AUC=6) IV Day 1 Repeat q 3 weeks x 6-10 cycles
- Regimen II - Uterine Carcinsarcoma Subjects; Regimen IV - Non-uterine Carcinsarcoma Subjects: Ifosfamide 1.6 g/m2 IV days 1, 2, 3 Mesna Paclitaxel 135 mg/m2 by 3-hour infusion on Day 1 Repeat q 3 weeks x 6-10 cycles. G-CSF Support: Filgrastim or Pegfilgrastim beginning Day 4-6
- Regimen III - Non-uterine Carcinsarcoma Subjects: Paclitaxel 175 mg/m2 IV over 3 hours Day 1 Carboplatin (AUC=6) IV Day 1 Repeat q 3 weeks x 6-10 cycles
Period: Overall Study
Arm/Group | Regimen I - Uterine Carcinsarcoma Subjects | Regimen II - Uterine Carcinsarcoma Subjects | Regimen III - Non-uterine Carcinsarcoma Subjects | Regimen IV - Non-uterine Carcinsarcoma Subjects
Started | 268 | 268 | 51 | 50
Completed | 142 | 145 | 27 | 25
Not Completed | 126 | 123 | 24 | 25
Not completed — Adverse Event | 28 | 23 | 4 | 9
Not completed — Death | 4 | 2 | 0 | 0
Not completed — Lack of Efficacy | 32 | 22 | 8 | 6
Not completed — Withdrawal by Subject | 14 | 10 | 4 | 3
Not completed — Medical Reason | 4 | 2 | 1 | 0
Not completed — Ineligible | 40 | 47 | 7 | 4
Not completed — Never Treated | 4 | 17 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen I - Uterine Carcinsarcoma Subjects | Regimen II - Uterine Carcinsarcoma Subjects | Regimen III - Non-uterine Carcinsarcoma Subjects | Regimen IV - Non-uterine Carcinsarcoma Subjects | Total
Number analyzed (Participants) | 228 | 221 | 44 | 46 | 539
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 3 | 0 | 0 | 3
  30-39 years | 1 | 1 | 2 | 0 | 4
  40-49 years | 12 | 8 | 3 | 2 | 25
  50-59 years | 46 | 45 | 12 | 18 | 121
  60-69 years | 111 | 111 | 15 | 15 | 252
  70-89 years | 58 | 53 | 12 | 11 | 134
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 221 | 44 | 46 | 539
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 2 | 3 | 17
  Not Hispanic or Latino | 215 | 206 | 42 | 40 | 503
  Unknown or Not Reported | 9 | 7 | 0 | 3 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
  Asian | 9 | 9 | 2 | 4 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 66 | 72 | 4 | 4 | 146
  White | 150 | 133 | 37 | 36 | 356
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 1 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Measured in months from randomization to last contact or death. Primary analysis was restricted to the eligible uterine carcinosarcoma cohort.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 115 months.
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Regimen I- Uterine Carcinsarcoma Subjects: Paclitaxel 175 mg/m2 IV over 3 hours Day 1 Carboplatin (AUC=6) IV Day 1 Repeat q 3 weeks x 6-10 cycles
Arm/Group | Regimen I- Uterine Carcinsarcoma Subjects | Regimen II - Uterine Carcinsarcoma Subjects
Number analyzed (Participants) | 228 | 221
months | 37.3 [25.7 to 49.0] | 29 [21.9 to 43.1]

2. Secondary Outcome: Duration of Progression-free Survival
Description: Measured in months from randomization to last contact or the earlier of the date of progression or death.
Time Frame: Approximately 9 years and 7 months
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regimen I - Uterine Carcinsarcoma Subjects | Regimen II - Uterine Carcinsarcoma Subjects | Regimen III - Non-uterine Carcinsarcoma Subjects | Regimen IV - Non-uterine Carcinsarcoma Subjects
Number analyzed (Participants) | 228 | 221 | 44 | 46
months | 16.3 [13.0 to 18.9] | 11.7 [10.1 to 17.3] | 14.6 [8.1 to 16.4] | 10.3 [8.5 to 19.0]

3. Secondary Outcome: Incidence of Adverse Events as Assessed by CTCAE Version 3.0
Description: Maximum grade experienced among all treated and eligible patients. The grades are described by severity. Grade 1 is the lowest (most mild) and Grade 5 being death (most severe). Adverse events were analyzed across cohorts since disease site was considered independent of AEs.
Time Frame: Patients were assessed for adverse events during active protocol treatment and up to 30 days after the last cycle of treatment on the protocol.
Population: Treated and Eligible subjects. Adverse events were analyzed across cohorts since disease site was considered independent of AEs.
Measure: Count of Participants; unit: Participants
Groups:
- Regimen I - Uterine and Non-Uterine Subjects: Paclitaxel 175 mg/m2 IV over 3 hours Day 1 Carboplatin (AUC=6) IV Day 1 Repeat q 3 weeks x 6-10 cycles
- Regimen II - All Uterine and Non-Uterine Subjects: Ifosfamide 1.6 g/m2 IV days 1, 2, 3 Mesna Paclitaxel 135 mg/m2 by 3-hour infusion on Day 1 Repeat q 3 weeks x 6-10 cycles. G-CSF Support: Filgrastim or Pegfilgrastim beginning Day 4-6
Arm/Group | Regimen I - Uterine and Non-Uterine Subjects | Regimen II - All Uterine and Non-Uterine Subjects
Number analyzed (Participants) | 268 | 247
Participants
  Grade 1 | 3 | 3
  Grade 2 | 22 | 80
  Grade 3 | 107 | 97
  Grade 4 | 130 | 61
  Grade 5 | 6 | 3

4. Secondary Outcome: Patient-Reported Quality of Life (QOL) - Baseline
Description: Patient reported quality of life was measured with the Treatment Outcome Index (TOI) of the Functional Assessment of Cancer Therapy for endometrial cancer (FACT-En TOI). The FACT-En TOI is a scale for assessing general QOL of endometrial cancer patients. The FACT-En TOI score ranges 0-120 with a large score suggesting better QOL. Quality of Life was analyzed across cohorts since disease site was considered independent of Quality of Life.
Time Frame: Baseline - Prior to study treatment
Population: Patients who provided baseline assessments.
Measure: Mean (Standard Error); unit: units on a scale (time point)
Groups:
- Regimen I - Uterine and Non-Uterine Subjects: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on day 1.
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Quality-of-Life Assessment: Ancillary studies
- Regimen II - Uterine and Non-Uterine Subjects: Patients receive ifosfamide IV over 1 hour on days 1-3 followed by paclitaxel as in Arm I.
  Ifosfamide: Given IV
  Paclitaxel: Given IV
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Regimen I - Uterine and Non-Uterine Subjects | Regimen II - Uterine and Non-Uterine Subjects
Number analyzed (Participants) | 205 | 184
units on a scale (time point) | 96.2 (1.1) | 97.5 (1.2)

5. Secondary Outcome: Patient Reported Quality of Life (QOL) - Post Baseline
Description: as for outcome 4
Time Frame: Prior to cycle 3, Prior to cycle 6, 30 weeks post cycle 1.
Population: Provided baseline and ≥ 1 follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale (time point)
Arm/Group | Regimen I - Uterine and Non-Uterine Subjects | Regimen II - Uterine and Non-Uterine Subjects
Number analyzed (Participants) | 205 | 184
units on a scale (time point)
  Pre-cycle 3 | 93.3 (0.9) | 93.3 (1.0)
  Pree-cycle 6 | 91.6 (1.1) | 91.6 (1.1)
  30 weeks post cycle 1 | 98.0 (1.1) | 97.6 (1.3)

6. Secondary Outcome: Patient Reported Peripheral Neuropathy Symptoms - Baseline
Description: Patient reported peripheral neuropathy symptoms was measured with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The FACT/GOG-Ntx subscale contains 11 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). . The Ntx score ranges 0-44 with a large score suggesting less peripheral neuropathy symptoms. Quality of Life was analyzed across cohorts since disease site was considered independent of Quality of Life.
Time Frame: Baseline (Pre cycle 1)
Population: Subjects who provided baseline assessment
Measure: Mean (Standard Error); unit: units on a scale-baseline
Arm/Group | Regimen I - Uterine and Non-Uterine Subjects | Regimen II - Uterine and Non-Uterine Subjects
Number analyzed (Participants) | 205 | 184
units on a scale-baseline | 40.2 (0.3) | 41.0 (0.3)

7. Secondary Outcome: Patient-reported Peripheral Neuropathy Symptoms - Post Baseline
Description: Patient reported peripheral neuropathy symptoms was measured with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The FACT/GOG-Ntx subscale contains 11 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). The Ntx score ranges 0-44 with a large score suggesting less peripheral neuropathy symptoms.Quality of Life was analyzed across cohorts since disease site was considered independent of Quality of Life.
Time Frame: Prior to cycle 3, Prior to cycle 6, 30 weeks post cycle 1
Population: Provided baseline and ≥ 1 follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Regimen I - Uterine and Non-Uterine Subjects | Regimen II - Uterine and Non-Uterine Subjects
Number analyzed (Participants) | 205 | 184
units on a scale
  Prior to cycle 3 | 37.2 (0.4) | 37.0 (0.5)
  Prior to cycle 6 | 34.1 (0.6) | 34.2 (0.6)
  30 weeks post cycle 1 | 34.8 (0.6) | 34.9 (0.6)

ADVERSE EVENTS:
Time Frame: Measured within 6 months of enrollment; through all cycles of chemotherapy and up to 30 days after the last cycle of chemotherapy. Up to 10 cycles of chemotherapy were allowed. Cycles were to be repeated every 3 weeks.
Description: Eligible and treated participants were affected if they experienced grade 1-5 adverse event. Adverse events were analyzed across cohorts since disease site was considered independent of AEs.
Groups:
- Regimen I - Uterine and Non-uterine Carcinosarcoma: Paclitaxel 175 mg/m2 IV over 3 hours Day 1 Carboplatin (AUC=6) IV Day 1 Repeat q 3 weeks x 6-10 cycles
- Regimen II - Uterine and Non-uterine Carcinsarcoma Subjects: Ifosfamide 1.6 g/m2 IV days 1, 2, 3 Mesna Paclitaxel 135 mg/m2 by 3-hour infusion on Day 1 Repeat q 3 weeks x 6-10 cycles. G-CSF Support: Filgrastim or Pegfilgrastim beginning Day 4-6
Arm/Group | Regimen I - Uterine and Non-uterine Carcinosarcoma | Regimen II - Uterine and Non-uterine Carcinsarcoma Subjects
All-Cause Mortality (participants affected / at risk) | 160/272 | 160/267
Serious Adverse Events (participants affected / at risk) | 80/268 | 68/247
Other Adverse Events (participants affected / at risk) | 268/268 | 244/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I - Uterine and Non-uterine Carcinosarcoma (N=268) | Regimen II - Uterine and Non-uterine Carcinsarcoma Subjects (N=247)
Neutrophils (Blood and lymphatic system disorders) | 32 | 12
Platelets (Blood and lymphatic system disorders) | 2 | 1
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 1
Cd4 Count (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 1 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 2
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1 | 1
Vasovagal Episode (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia - Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 | 1
Hypertension (Cardiac disorders) | 1 | 0
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 1 | 0
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Cardipulmonary Arrest (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1 | 1
Death No Ctcae Term - Death Nos (General disorders) | 2 | 0
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 1 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Ulcer,gi - Esophagus (Gastrointestinal disorders) | 0 | 1
Perforation, Gi - Colon (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Dehydration (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Wound (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1 | 1
Febrile Neutropenia (Infections and infestations) | 3 | 2
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Blood (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 1 | 2
Inf W/Gr 3 Or 4 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1 | 1
Inf Unknown Anc: Foreign Body (Infections and infestations) | 0 | 1
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 1
Inf Unknown Anc: Colon (Infections and infestations) | 1 | 0
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Vulva (Infections and infestations) | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Apnea (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Speech Impairment (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 1 | 0
Confusion (Nervous system disorders) | 0 | 5
Dizziness (Nervous system disorders) | 0 | 1
Pain - Other (General disorders) | 1 | 1
Pain: Pelvis (General disorders) | 0 | 1
Pain: Chest /Thorax Nos (General disorders) | 0 | 3
Pain: Head/Headache (General disorders) | 1 | 0
Pain: Extremity-Limb (General disorders) | 1 | 0
Pain: Back (General disorders) | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 3 | 0
Pain: Cardiac/ Heart (General disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 3
Cytokine Release Syndrome (General disorders) | 2 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 2 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 | 4
Death No Ctcae Term - Sudden Death (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen I - Uterine and Non-uterine Carcinosarcoma (N=268) | Regimen II - Uterine and Non-uterine Carcinsarcoma Subjects (N=247)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 19 | 11
Rhinitis (Immune system disorders) | 6 | 12
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 | 2
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 8 | 4
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 2 | 0
Neutrophils (Blood and lymphatic system disorders) | 245 | 116
Platelets (Blood and lymphatic system disorders) | 178 | 137
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 7 | 9
Bone Marrow Cellularity (Blood and lymphatic system disorders) | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 239 | 164
Lymphopenia (Blood and lymphatic system disorders) | 18 | 26
Hemoglobin (Blood and lymphatic system disorders) | 249 | 232
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 3 | 1
Conduction Abnml: Conduction Abnormality Nos (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 8 | 8
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 1
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 4 | 6
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 2
Hypertension (Cardiac disorders) | 26 | 25
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 1 | 0
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 2
Cardiac General - Other (Cardiac disorders) | 1 | 1
Cardiac Troponin I (Ctni) (Cardiac disorders) | 0 | 1
Cardiac Troponin T (Ctnt) (Cardiac disorders) | 1 | 0
Hypotension (Cardiac disorders) | 12 | 8
Inr (Vascular disorders) | 3 | 4
Coagulopathy - Other (Vascular disorders) | 1 | 0
Ptt (Vascular disorders) | 1 | 2
Constitutional Symptoms - Other (General disorders) | 2 | 4
Sweating (General disorders) | 5 | 8
Weight Gain (General disorders) | 7 | 14
Patient Odor (General disorders) | 0 | 1
Fever (General disorders) | 7 | 16
Weight Loss (General disorders) | 14 | 19
Rigors/Chills (General disorders) | 8 | 7
Fatigue (General disorders) | 192 | 177
Insomnia (General disorders) | 43 | 35
Nail Changes (Skin and subcutaneous tissue disorders) | 12 | 15
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 | 2
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 190 | 171
Induration (Skin and subcutaneous tissue disorders) | 0 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 8 | 6
Bruising (Skin and subcutaneous tissue disorders) | 4 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 24 | 23
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 8
Decubitus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Flushing (Skin and subcutaneous tissue disorders) | 1 | 5
Hand-Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 13
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 2
Hot Flashes (Endocrine disorders) | 17 | 19
Diabetes (Endocrine disorders) | 1 | 3
Hypothyroidism (Endocrine disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Ulcer,gi - Duodenum (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 3
Esophagitis (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 5 | 3
Heartburn (Gastrointestinal disorders) | 21 | 20
Dental: Teeth (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 4
Dysphagia (Gastrointestinal disorders) | 4 | 2
Distention (Gastrointestinal disorders) | 7 | 8
Taste Alteration (Gastrointestinal disorders) | 25 | 42
Incontinence, Anal (Gastrointestinal disorders) | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 4 | 5
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 5 | 14
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 2
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 10 | 12
Mucositis (Clinical Exam) - Larynx (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 51 | 64
Anorexia (Gastrointestinal disorders) | 61 | 67
Dehydration (Gastrointestinal disorders) | 18 | 18
Constipation (Gastrointestinal disorders) | 129 | 119
Nausea (Gastrointestinal disorders) | 132 | 131
Gastrointestinal - Other (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 77 | 55
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 1 | 14
Hemorrhage, Gu - Vagina (Vascular disorders) | 7 | 4
Hemorrhage, Gu - Urethra (Vascular disorders) | 1 | 0
Hemorrhage, Gi - Rectum (Vascular disorders) | 2 | 3
Hemorrhage, Gi - Peritoneal Cavity (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 0 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 6 | 7
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage, Gu - Uterus (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 1 | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 1 | 8
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Wound (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Dental-Tooth (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 5 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Pleura (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Lymphatic (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 5 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1 | 0
Febrile Neutropenia (Infections and infestations) | 5 | 1
Inf Unknown Anc: Bone (Osteomyelitis) (Infections and infestations) | 0 | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 1 | 0
Viral Hepatitis (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 15 | 17
Inf Unknown Anc: Blood (Infections and infestations) | 0 | 1
Infection - Other (Infections and infestations) | 5 | 4
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 0 | 2
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 2
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 2 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 1
Inf Unknown Anc: Bronchus (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc:peritoneal Cavity (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 5 | 6
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1 | 2
Inf Unknown Anc: Wound (Infections and infestations) | 2 | 1
Inf Unknown Anc: Foreign Body (Infections and infestations) | 1 | 0
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 1 | 1
Inf W/Gr 3 Or 4 Anc: Vagina (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Pelvis Nos (Infections and infestations) | 1 | 1
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 2
Inf W/Gr 3 Or 4 Anc: Bronchus (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2 | 3
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 3 | 2
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1 | 1
Edema: Limb (Blood and lymphatic system disorders) | 43 | 40
Edema: Head And Neck (Blood and lymphatic system disorders) | 1 | 2
Ast (Metabolism and nutrition disorders) | 20 | 19
Gfr (Metabolism and nutrition disorders) | 5 | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 8 | 4
Proteinuria (Metabolism and nutrition disorders) | 1 | 13
Creatinine (Metabolism and nutrition disorders) | 30 | 34
Hypoalbuminemia (Metabolism and nutrition disorders) | 41 | 46
Ggt (Metabolism and nutrition disorders) | 0 | 2
Alt (Metabolism and nutrition disorders) | 14 | 21
Alkaline Phosphatase (Metabolism and nutrition disorders) | 23 | 50
Bilirubin (Metabolism and nutrition disorders) | 5 | 3
Lipase (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 13 | 24
Hyponatremia (Metabolism and nutrition disorders) | 38 | 25
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 3 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 22 | 36
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 62 | 64
Hypokalemia (Metabolism and nutrition disorders) | 48 | 49
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 8
Hypercalcemia (Metabolism and nutrition disorders) | 14 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 69 | 18
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 4 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Gait/Walking (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 5
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 24 | 15
Muscle Weakness - Trunk (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 4 | 5
Syncope (Nervous system disorders) | 4 | 5
Involuntary Movement (Nervous system disorders) | 3 | 4
Pyramidal Tract Dysfunction (Nervous system disorders) | 0 | 1
Psychosis (Nervous system disorders) | 1 | 1
Myelitis (Nervous system disorders) | 0 | 2
Neurology - Other (Nervous system disorders) | 2 | 2
Mental Status (Nervous system disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 22 | 31
Mood Alteration - Anxiety (Nervous system disorders) | 27 | 27
Mood Alteration - Agitation (Nervous system disorders) | 4 | 2
Tremor (Nervous system disorders) | 1 | 3
Speech Impairment (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 2 | 2
Personality (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 4
Cognitive Disturbance (Nervous system disorders) | 4 | 2
Cns Ischemia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 4 | 11
Memory Impairment (Nervous system disorders) | 11 | 10
Dizziness (Nervous system disorders) | 33 | 27
Neuropathy,cranial - Cn Vii Motor-Face (Nervous system disorders) | 1 | 0
Neuropathy-Sensory (Nervous system disorders) | 178 | 158
Neuropathy-Motor (Nervous system disorders) | 5 | 6
Ocular/Visual - Other (Eye disorders) | 1 | 2
Watery Eye (Eye disorders) | 2 | 5
Dry Eye (Eye disorders) | 3 | 4
Cataract (Eye disorders) | 2 | 2
Photophobia (Eye disorders) | 1 | 0
Flashing Lights/Floaters (Eye disorders) | 3 | 4
Blurred Vision (Eye disorders) | 18 | 13
Keratitis (Eye disorders) | 1 | 0
Eyelid Dysfunction (Eye disorders) | 0 | 1
Pain - Other (General disorders) | 9 | 9
Pain: Urethra (General disorders) | 4 | 4
Pain: Perineum (General disorders) | 1 | 0
Pain: Pelvis (General disorders) | 4 | 2
Pain: Breast (General disorders) | 1 | 1
Pain: Vagina (General disorders) | 1 | 1
Pain: Chest /Thorax Nos (General disorders) | 7 | 10
Pain: Chest Wall (General disorders) | 1 | 4
Pain: Throat/Pharynx/Larynx (General disorders) | 3 | 5
Pain: Eye (General disorders) | 0 | 1
Pain: Head/Headache (General disorders) | 30 | 34
Pain: Neck (General disorders) | 2 | 2
Pain: Intestine (General disorders) | 1 | 0
Pain: Extremity-Limb (General disorders) | 32 | 23
Pain: Buttock (General disorders) | 0 | 1
Pain: Back (General disorders) | 25 | 35
Pain: Joint (General disorders) | 58 | 41
Pain: Bone (General disorders) | 20 | 45
Pain: Bladder (General disorders) | 2 | 2
Pain: Pain Nos (General disorders) | 8 | 1
Pain: Stomach (General disorders) | 4 | 2
Pain: Oral Cavity (General disorders) | 1 | 1
Pain: Esophagus (General disorders) | 1 | 0
Pain: Dental/Teeth/Peridontal (General disorders) | 3 | 0
Pain: Abdominal Pain Nos (General disorders) | 47 | 56
Pain: Scalp (General disorders) | 1 | 1
Pain: Oral - Gums (General disorders) | 0 | 1
Pain: Lip (General disorders) | 1 | 0
Pain: Middle Ear (General disorders) | 0 | 1
Pain: External Ear (General disorders) | 4 | 0
Pain: Cardiac/ Heart (General disorders) | 1 | 2
Pain: Face (General disorders) | 2 | 0
Pain: Muscle (General disorders) | 46 | 41
Pain: Anus (General disorders) | 1 | 2
Pain: Neuralgia (General disorders) | 0 | 1
Pain: Sinus (General disorders) | 0 | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Prolonged Intubation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 37
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 55 | 48
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 | 13
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Leak, Gu - Vagina (Renal and urinary disorders) | 0 | 1
Leak, Gu - Bladder (Renal and urinary disorders) | 1 | 1
Cystitis (Renal and urinary disorders) | 3 | 4
Urinary Color Change (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 2
Urinary Electrolyte Wasting (Renal and urinary disorders) | 0 | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 2
Incontinence, Urinary (Renal and urinary disorders) | 15 | 11
Fistula, Gu - Vagina (Renal and urinary disorders) | 0 | 1
Bladder Spasm (Renal and urinary disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 7 | 9
Urinary Frequency (Renal and urinary disorders) | 25 | 16
Nipple/Areolar (Reproductive system and breast disorders) | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 3 | 2
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 0 | 1
Vaginitis (Reproductive system and breast disorders) | 3 | 0
Vaginal Mucositis (Reproductive system and breast disorders) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 4 | 10
Syndromes - Other (General disorders) | 1 | 1
Cytokine Release Syndrome (General disorders) | 1 | 0
Flu-Like Syndrome (General disorders) | 3 | 1
Vascular - Other (Vascular disorders) | 1 | 2
Vein Injury - Jugular (Vascular disorders) | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 2 | 3
Thrombosis/Thrombus/Embolism (Vascular disorders) | 15 | 6
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT00954174/Prot_SAP_000.pdf